CLINICAL TRIAL: NCT03820427
Title: Evaluation of Novel Lung Function Parameters in Patients With Bronchial Asthma
Status: Completed | Type: Observational
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Dr. Frederik Trinkmann, Principal Investigator, Universitätsmedizin Mannheim
Other Study IDs: MBW-asthma
Record Dates: First submitted 2019-01-22; First posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Bronchial Asthma; Pulmonary Healthy Controls
MeSH Terms: conditions — Asthma | interventions — Plethysmography, Whole Body

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- bronchial asthma: Patients with known or suspected asthma.
  Interventions: Diagnostic Test: impulse oscillometry; Diagnostic Test: multiple breath washout test; Diagnostic Test: body plethysmography
- pulmonary healthy controls: Patients without known or suspected pulmonary disease
  Interventions: Diagnostic Test: impulse oscillometry; Diagnostic Test: multiple breath washout test; Diagnostic Test: body plethysmography

INTERVENTIONS:
Diagnostic Test: impulse oscillometry — impulse oscillometry
Diagnostic Test: multiple breath washout test — multiple breath washout test
Diagnostic Test: body plethysmography — body plethysmography

SUMMARY:
Current guideline-based criteria defining bronchial asthma do not always meet the challenges set by the complex pathophysiology of the disease. The investigators therefore aimed to evaluate novel or not widely used functional diagnostic approaches for the detection and therapeutic monitoring of patients with asthma.

ELIGIBILITY:
Inclusion Criteria:

* known or suspected bronchial asthma
* known or suspected obstructive ventilation disorder
* pulmonary healthy controls

Exclusion Criteria:

* pregnancy
* inability to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with indication for routine lung function testing
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Global ventilation heterogeneity | 30 minutes
  lung clearance index (LCI) derived from sulphur hexafluoride multiple breath washout
Local ventilation heterogeneity | 30 minutes
  Sacin, Scond (Phase III slopes) derived from sulphur hexafluoride multiple breath washout

IPD SHARING:
Plan to Share IPD: No